CLINICAL TRIAL: NCT05165628
Title: A Randomised, Controlled, Phase 1 Study to Investigate Safety, Tolerability and Efficacy of CYP-006TK in Adults with Diabetic Foot Ulcers
Brief Title: Safety, Tolerability and Efficacy of CYP-006TK in Adults with Diabetic Foot Ulcers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cynata Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CYP-DFU-P1-01
Record Dates: First submitted 2021-10-18; First posted 2021-12-21 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Foot Ulcer; Cutaneous Ulcer
MeSH Terms: conditions — Diabetic Foot; Skin Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 - CYP-006TK (Experimental): Participants will receive CYP-006TK dressings
  Interventions: Combination Product: CYP-006TK
- Group 2 - Standard of Care (No Intervention): Participants will continue to be treated as per local standard of care

INTERVENTIONS:
Combination Product: CYP-006TK — CYP-006TK is allogenic mesenchymoangioblast-derived mesenchymal stem cells (MCA-derived MSCs) or Cymerus™ MSCs, seeded onto a heptylamine plasma polymer-coated silicone dressing
  Arms: Group 1 - CYP-006TK

SUMMARY:
Design: A randomised, controlled, prospective trial. Participants will be patients with non-healing diabetic foot ulcers.

The study will aim to recruit 15 participants per study group (30 participants in total). Participants will be randomly allocated to one of two treatment groups:

* Group 1: CYP-006TK
* Group 2: Standard care This will be an open label study with respect to treatment allocation. However, the person reviewing images of the study ulcers to assess healing will be blind to the participant's treatment allocation.

Participants assigned to Group 1 will be treated with CYP-0006TK dressings on 8 occasions over 4 weeks. The dressings will be changed every 3 or 4 days. After the first 4 weeks, participants in Group 1 will revert to standard care for the rest of the study. Participants assigned to Group 2 will have their ulcer treated with standard care throughout the study.

Participants will attend a total of 16 scheduled visits over 24 weeks. There will be a mixture of on-site (hospital/clinic) visits, and home visits. The study will end 24 weeks after the initiation of treatment, unless the study ulcer is completely headed before then.

ELIGIBILITY:
Inclusion Criteria:

1. Adults at least 18 years of age up to 80 years of age, inclusive.
2. Have a current diagnosis of diabetes mellitus (DM)
3. With at least one non-healing cutaneous ulcer on the foot or the lower legs
4. With ankle brachial index (ABI) ≥ 0.4 and/or toe pressure >30 mmHg on the limb with the study ulcer.
5. Participant co-morbidities are adequately managed, and the participant has a life expectancy of at least 6 months as determined by the Investigator based on medical history, physical examination, vital signs, or clinical laboratory tests, etc.
6. A negative pregnancy test, (i.e. for female participants with childbearing potential).
7. Willing to comply with birth control measures, to prevent female participants becoming pregnant for six months following administration of the study treatment.
8. Able to follow the Investigator's instruction on ulcer care (in the opinion of the Investigator).
9. Agrees to provide written informed consent.

Exclusion Criteria:

1. Planned vascular surgery, angioplasty, thrombolysis or amputation of the affected limb in the next six months.
2. Pregnant or breastfeeding.
3. Active infection in the study ulcer.
4. Any sign of osteomyelitis associated with the study ulcer.
5. Study ulcer extends to bone or periosteum (ulcers that reach a ligament, joint capsule, fascia, or tendon are not excluded).
6. Study ulcer requires daily dressing changes.
7. Known autoimmune disease other than diabetes, including but not limited to lupus erythematosus, multiple sclerosis which are considered as clinically significant by PI and/or Medical Monitor.
8. Treatment with systemic immunosuppressants within 90 days of screening.
9. Active malignancy or history of malignancy within five years prior to screening (with the exception of a past history of basal or squamous cell carcinomas).
10. Serum GGT, AST or ALT > 5 × upper limit of the normal range (ULN).
11. . Known history of HIV infection
12. Prior administration of any cell-based treatment to the limb affected by the study ulcer.
13. Received any investigational research agent within 60 days or within five half-lives of the last treatment (if the half-life of the investigational agent is known to be longer than 12 days) prior to the planned initiation of study treatment.
14. Any other medical condition or laboratory abnormality judged as clinically significant by the Investigator or study Medical Monitor which could confound the evaluation of the trial treatment.
15. With history of sensitivity to materials of bovine, porcine origin, or human serum albumin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (TEAEs) | 24 weeks
Incidence of changes from baseline in haematology, biochemistry, and urinalysis parameters. | 24 weeks
  Results will be summarised by individual and by treatment group using descriptive statistics.

SECONDARY OUTCOMES:
Percentage of area change of study ulcer from baseline to weeks 12 and 24 | 12 and 24 weeks
Number of days to complete ulcer healing | 12 and 24 weeks
Number of days to 50% ulcer healing | 12 and 24 weeks
Percentage change in ulcer volume from baseline to weeks 12 and 24 | 12 and 24 weeks
Changes from baseline in ulcer pain assessed using a Numeric Rating Scale | 12 and 24 weeks
Number clinic/home care visits across groups | 12 and 24 weeks
Differences across groups on ulcer dressing products used | 12 and 24 weeks
Changes from baseline in Quality of Life assessed using the Cardiff Wound Impact Schedule | 12 and 24 weeks
Duration of clinic/home care visits across groups | 12 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jolanta Airey, MD, Study Director — Cynata Therapeutics Limited
Locations (4):
- Australia (4):
  - Central Adelaide Local Health Network, Adelaide, South Australia
  - Fiona Stanley Hospital, Perth, Western Australia
  - Royal Perth Hospital, Perth, Western Australia
  - Sir Charles Gairdner Hospital, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No